CLINICAL TRIAL: NCT01125709
Title: Comparative Study of Clinical Endpoint in DMD: HHM vs. CQMS
Brief Title: Comparative Study of Clinical Endpoint in DMD: Handheld Myometry (HHM) Versus CINRG Quantitative Measurement System (CQMS)
Status: Completed | Type: Observational
Sponsor: Cooperative International Neuromuscular Research Group (Network)
Collaborators: Muscular Dystrophy Association (Other); Children's National Research Institute (Other); Washington University School of Medicine (Other); Royal Children's Hospital (Other); Sydney Children's Hospitals Network (Other); Fondazione Serena Onlus - Centro Clinico NeMO Milano (Other); Carolinas Medical Center (Other)
Responsible Party: Tina Duong, MPT, Children's National Medical Center, Children's Research Institute
Other Study IDs: CNMC0609
Record Dates: First submitted 2010-05-17; First posted 2010-05-18 (Estimated); Last update posted 2013-01-11 (Estimated); Status verified 2013-01

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Neuromuscular disease; Duchenne; Muscular Dystrophy; DMD; Strength assessment; CINRG Quantitative Measurement System; CQMS; Hand Held Myometry; HHM
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Neuromuscular Diseases; Muscular Dystrophies

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of the proposed research is to compare two commonly used pediatric strength testing measures: handheld myometry (HHM) and CINRG Quantitative Measurement System (CQMS), with the goal of identifying a sensitive and valid tool for measuring muscle strength in children with DMD. The data obtained from this study will be used to make recommendations for strength measurement endpoints in prospective muscular dystrophy trials and provide more reliable and accurate recommendations in the clinic for strength assessment. This study will be performed at six participating sites in the Cooperative International Neuromuscular Research Group (CINRG).

DETAILED DESCRIPTION:
We propose to compare the reliability of CQMS vs. HHM in the DMD population. The importance of this study is to be able to compare the results of clinical trials done by different networks using distinct strength endpoints. If results indicate a distinct difference in reliability of one tool over the other, a standardized tool could be established for research groups throughout the world to interpret strength in the context of clinical trials. If the results indicate minor differences then it would be possible to interpret and compare/contrast strength measurements used in different studies.

Understanding the relationship between the HHM vs CQMS will help us examine other surrogate measures capable of predicting functionality that are based on strength measurements.

ELIGIBILITY:
Participants should meet the following criteria:

1. Confirmed clinical and molecular diagnosis of DMD
2. 6- 18 years of age
3. Ability to follow 2 step instructions
4. Ability to transfer to and from the wheelchair-mat with moderate assistance defined as no greater than 75% assistance.
5. Signed informed consent of parental or legal guardian(s) is required for participants. Assent from children 7-18 years old may also required.

Exclusion Criteria:

Participants must confirm:

1. No Surgical procedures were performed ≤ 8 weeks before study procedures.
2. No musculoskeletal injuries were experienced ≤ 8 weeks before study procedures.
3. Investigator assessment that patient or parent/legal guardian are not willing or able to comply with study procedures.

Ages: 6 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants will be selected from participating CINRG institution's neuromuscular clinics.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Compare the inter and intra rater reliability of HHM and CQMS by measuring Elbow and Knee Flexor/Extensor Strength in children ages 6-18 diagnosed with DMD tested by experienced clinical evaluators in both HHM and CQMS. | two-day visit
  Muscle groups will be tested in a standardized order 1. Knee extension 2. Knee flexion 3. Elbow Flexion 4. Elbow extension with all tests sequencing following a right to left pattern. This will reduce assessment bias and the impact of muscle fatigue per muscle group. Study participants are randomized to two different sequences of four assessments, one sequence performed on one testing day (Visit 1) and another on a different testing day (Visit 2).

CONTACTS AND LOCATIONS:
Overall Officials: Tina T Duong, MPT, Principal Investigator — Children's National Research Institute
Locations (5):
- United States (3):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Washington University - St. Louis, St Louis, Missouri
  - Carolinas Medical Center, Charlotte, North Carolina
- Royal Children's Hospital, Parkville, Victoria, Australia
- Centro Clinico Nemo, Milan, Italy

REFERENCES:
- See also: CINRG website where all current and completed protocols are listed. — http://www.cinrgresearch.org